CLINICAL TRIAL: NCT02710461
Title: Acute Effects of Grape and Pomegranate Polyphenols as Modulators of Metabolic Syndrome in Humans
Brief Title: Grape and Pomegranate Polyphenols in Postprandial Glucose and Related Parameters
Acronym: POME-GRAPE-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Jara Pérez-Jiménez, PhD, National Research Council, Spain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AGL2014-55102-JIN_1
Record Dates: First submitted 2016-03-12; First posted 2016-03-16 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Subjects With Abdominal Obesity
Keywords: Polyphenols; Grape; Pomegranate; Metabolic syndrome; Abdominal obesity; Postprandial glucose; Insulin resistance
MeSH Terms: conditions — Metabolic Syndrome; Obesity, Abdominal; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects with abdominal obesity (Experimental): Intervention with grape pomace and pomegranate pomace
  Interventions: Dietary Supplement: Mixture of grape pomace and pomegranate pomace

INTERVENTIONS:
Dietary Supplement: Mixture of grape pomace and pomegranate pomace — Oral Glucose Tolerance Test
Dietary Supplement: Mixture of grape pomace and pomegranate pomace — Oral Glucose Tolerance Test right after taking the mixture of grape and pomegranate polyphenols
Dietary Supplement: Mixture of grape pomace and pomegranate pomace — Oral Glucose Tolerance Test ten hours after taking the mixture of grape and pomegranate polyphenols

SUMMARY:
The aim of this is study is to evaluate the acute effect of grape and pomegranate polyphenols in the modulation of markers of metabolic syndrome. Most of the previous works about polyphenols have only considered a fraction of polyphenols, i.e., extractable polyphenols. As a consequence, an important amount of dietary polyphenols, the so-called non-extractable polyphenols are ignored. In contrast, the effect of both extractable and non-extractable polyphenols will be considered in this study. Furthermore, the effect of both polyphenols as present in the food matrix and metabolites derived from microbial fermentation will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal perimeter ≥102 cm. for male participants and ≥88 cm for female participants.
* Subjects presenting some or several of these characteristics will be prioritized:

Fasting glucose values between 110-128 mg/dL. Triglycerides = 150-195 mg/dL. HDL-cholesterol: < 50 mg/dL men, < 40 mg/dL women. Blood pressure: systolic > 130 mm Hg; diastolic > 85 mm Hg.

Exclusion Criteria:

* Subjects taking drugs for hyperglycaemia, hypertension or hypercholesterolaemia.
* Volunteers participating in other studies or weight loss plans.
* Pregnant or breastfeeding women.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose | 0-120 min.
  Changes in blood glucose response in treatments B and C will be compared with the baseline results obtained in treatment A. This will be evaluated by area under the curve (AUC) 0-120 min after an Oral Glucose Tolerance Test (OGTT)

SECONDARY OUTCOMES:
Postprandial insulin | 0-120 min.
  Changes in blood insulin response in treatments B and C will be compared with the baseline results obtained in treatment A. This will be evaluated by area under the curve (AUC) 0-120 min after an Oral Glucose Tolerance Test (OGTT)
Postprandial uric acid | 0-120 min.
  Changes in blood uric acid response in treatments B and C will be compared with the baseline results obtained in treatment A. This will be evaluated by area under the curve (AUC) 0-120 min after an Oral Glucose Tolerance Test (OGTT)
Polyphenol metabolites | 0-180 min.
  Urinary polyphenol metabolites will be determined in samples collected in the period 0-180 min. of each intervention.
Urinary uric acid | 0-180 min.
  Urinary uric acid will be determined in samples collected in the period 0-180 min. of each intervention.
Satiety | 120 min.
  A satiety test, including 10 items, will be provided at different time points during the period 0-120 min. of each intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Food Science, Technology and Nutrition, National Research Council (ICTAN-CSIC), Madrid, Madrid, Spain